CLINICAL TRIAL: NCT07126197
Title: Using Lymphovenous Bypass to Alleviate Diabetic Peripheral Neuropathy
Acronym: LVB ease DPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202503048RINA; 114-R0011 (Other Grant/Funding Number: National Taiwan University Hospital)
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathy (DPN); Diabetic Peripheral Neuropathic Pain (DPNP); Diabetic Foot Ulcer
Keywords: lymphaticovenular anastomosis; lymphovenous bypass
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The protocol begins with patient recruitment from two clinics, followed by a joint DM co-care evaluation. Eligible patients who consent undergo baseline data collection, including demographics, lab work, and neuropathy tests (Sudoscan, HRV, QST, MNSI, DN4).
  Participants allocated to DPN, DPNP, and DFU subgroups will undergo a key step involves a lymphovenous bypass surgery (with/without) and a biopsy to assess Intra-Epidermal Nerve Fiber (IENF) density.
  The study includes follow-up visits at 6 and 12 months for repeated neuropathy evaluations. Another skin biopsy for IENF density is also performed at the 12-month check-up. The final stage involves a comparative analysis of the data collected from all groups to assess outcomes.
  Exclusion criteria include patients with amputations, specific drug prescriptions, and severe peripheral artery disease (ABI ≤ 0.9).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients having DPN(P) with/without DFUs undergo lymphovenous bypass (Experimental): Patients having DPN(P) with/without DFUs undergo lymphovenous bypass and biopsy at foot dorsum. DPN n = 10, DPNP n = 10, DFU n = 20
  Interventions: Procedure: lymphovenous bypass at diseased foot dorsum

INTERVENTIONS:
Procedure: lymphovenous bypass at diseased foot dorsum — A lymphovenous bypass procedure using a lymphangiography dye (Patent Blue V or indocyanine green), 0.2 mL was injected into the skin at the toe webspaces preoperatively. 8,13,14 The paths of lymphatic vessels were traced. On the foot dorsum of the affected limb, a horizontal incision of 2-3 cm was made close to the lymphatic vessel's pathway. Under the surgical microscope, suitable lymphatic and venous vessels were identified, usually located above the deep fascia (on the superficial side, ensuring that the extensor hallucis longus tendon remains unexposed). The coaptation between the lymphatic vessels and venules followed the same principles as those for vascular anastomosis by using higher magnification under the surgical microscope (approximately 20×), finer microsurgical instruments, and 11- or 12-0 nylon sutures.

SUMMARY:
Diabetes is a metabolic disease characterized by high blood sugar levels due to a lack of insulin. Long-term metabolic disorders can cause structural and functional changes in many organs, mainly affecting the vascular system, and leading to complications in the eyes, kidneys, and nervous system. Diabetic Peripheral Neuropathy (DPN) is a common complication, affecting about 50% of patients. According to the Chinese Diabetes Association, DPN is diagnosed when diabetic patients exhibit signs of peripheral nerve dysfunction, as determined by physical examination or electrophysiological testing, after excluding other causes. The prevalence of DPN in diabetic patients is generally over 30%, with 20-30% experiencing significant pain and mobility issues, severely affecting quality of life and increasing the risk of amputation. Prevention and control rely on strict blood sugar management and lifestyle adjustments, as no medication or surgical intervention can cure DPN.

The lymphatic system plays an immunological role in regulating immune cell migration and inflammatory responses. Supermicrosurgical lymphovenous bypass (LVB) has become a routine treatment for lymphedema, allowing high-pressure lymph fluid to drain into non-occluded deep venous systems, alleviating lymphedema, restoring TH1 and TH2 balance, reducing oxidative stress, and enhancing antioxidant capacity. LVB may delay DPN progression, alleviate pain (DPNP), and promote diabetic foot ulcer healing. In our clinical experience, a patient with Charcot's neuroarthropathy and chronic plantar ulcers underwent LVB alongside wound care. Five years of follow-up showed complete wound healing without further amputation, despite poor HbA1c control. Thus, we aim to further accumulate clinical experience and data, study histological changes, and confirm the benefits of this surgery to help similar patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 80 years old.
* Gender: no distinction.
* Patients diagnosed with diabetic peripheral neuropathy, with or without diabetic foot ulcers, but there will be different groups.
* Patients can cooperate with doctors' orders as much as possible.
* Wound care that requires regular wound cleaning and dressing changes by nursing staff.
* Agree to join this study and sign the consent form.

Exclusion Criteria:

* Patients with autoimmune diseases, such as systemic lupus erythematosus.
* Patients with organ failure, such as heart, lung, kidney, and liver failure.
* Patients with diabetic foot ulcers and severe infections that require amputation of the forefoot.
* Patients with significant cognitive impairment or insufficient consciousness and unable to understand the purpose of the plan.
* Under 20 years old and over 80 years old.
* Patients receiving palliative care.
* Pregnant women.
* Patients whose physical condition cannot accept general anesthesia or surgery.
* Patients who are allergic to Patent Blue V or Gentian Violet injection for lymphatic visualization.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sudoscan | Preoperative, Postoperative 6 and 12 months
  Sudoscan is a non-invasive medical device that assesses sweat gland function, specifically measuring sweat chloride concentrations in the palms and soles. This provides an indirect measure of small fiber neuropathy, as these nerve fibers innervate the sweat glands. The test involves placing a patient's hands and feet on electrodes, and a low-voltage electrical current is passed through the skin. The device then calculates electrochemical skin conductance (ESC). Abnormal ESC values can indicate autonomic neuropathy, a common complication of conditions like diabetes, affecting nerves responsible for involuntary bodily functions.
Heart Rate Variability (HRV) | Preoperative, Postoperative 6 and 12 months
  HRV measures the variation in time between consecutive heartbeats. It reflects the balance and responsiveness of the autonomic nervous system, specifically the sympathetic ("fight or flight") and parasympathetic ("rest and digest") branches. A higher HRV generally indicates a more flexible and adaptable nervous system, associated with better health and stress resilience. A lower HRV can signal chronic stress, fatigue, or underlying health issues. It is a non-invasive tool used to assess cardiovascular health and monitor recovery.
Quantitative Sensory Testing (QST) | Preoperative, Postoperative 6 and 12 months
  QST is a non-invasive method for assessing the function of sensory nerve fibers. It measures a person's ability to feel and respond to various stimuli, such as temperature (cold and warm detection thresholds) and vibration. By applying controlled stimuli and recording the patient's perception, clinicians can identify and quantify sensory deficits. QST helps diagnose and monitor conditions affecting the peripheral nervous system, such as diabetic neuropathy, and can be used to track disease progression or the effectiveness of treatments.
Michigan Neuropathy Screening Instrument (MNSI) | Preoperative, Postoperative 6 and 12 months
  The MNSI is a two-part tool for screening for diabetic peripheral neuropathy. The first part is a 15-item patient questionnaire that asks about common neuropathic symptoms like numbness, burning pain, and muscle cramps. The second part is a physical examination conducted by a healthcare professional. This exam includes a visual inspection of the feet for deformities or ulcers, an assessment of ankle reflexes, and a crucial test of vibratory sensation using a tuning fork. The MNSI provides a quick, cost-effective way to identify patients who may need further diagnostic evaluation for neuropathy.
DN4 (Douleur Neuropathique en 4 Questions) | Preoperative, Postoperative 6 and 12 months
  The DN4 is a questionnaire specifically designed to identify neuropathic pain, which is a common and often debilitating symptom of diabetic neuropathy. It consists of 10 questions divided into two sections. The first part involves interviewing the patient about their pain characteristics, asking if they experience sensations like burning, cold, electric shocks, tingling, or numbness. The second part is a brief physical examination where the clinician checks for reduced sensation to touch or pinprick and if light brushing causes pain. A score of 4 or more out of 10 suggests the presence of neuropathic pain.
Intra-Epidermal Nerve Fiber (IENF) density | Preoperative and Postoperative 12 months
  IENF density is a quantitative measure used to assess the health of small nerve fibers. It is determined by counting the number of nerve fibers within a specific length of the epidermis, typically from a small skin biopsy. A reduction in IENF density is a key marker of small fiber neuropathy, an early sign of conditions like diabetic neuropathy. Because these fibers are among the first to be damaged, measuring IENF density is considered a highly sensitive and objective method for diagnosing and monitoring the progression of the disease.

IPD SHARING:
Plan to Share IPD: No